CLINICAL TRIAL: NCT00945308
Title: Effectiveness of Intracoronary Injection of Eptifibatide as Adjunctive Antiplatelet Therapy in Primary Coronary Intervention in Patients With ST Segment Elevation Acute Myocardial Infarction.
Brief Title: Effectiveness of Intracoronary Injection of Eptifibatide in Primary Coronary Intervention in STEMI Patients
Acronym: ICE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Alberto Hendler MD, Assaf harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 97/09
Record Dates: First submitted 2009-07-08; First posted 2009-07-24 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2009-07

CONDITIONS: Acute Myocardial Infarction
Keywords: Primary PCI; Acute myocardial infarction; Myocardial blush; Primary coronary intervention in acute myocardial infarction; focusing on the effect of the study drug on the immediate TIMI; flow at the infarct related artery and on the myocardial; perfusion evaluated by the TIMI myocardial perfusion grade or; blush
MeSH Terms: conditions — Blushing | interventions — Eptifibatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eptifibatide (intracoronary) (Active Comparator)
  Interventions: Drug: Eptifibatide
- Eptifibatide (intravenous) (Active Comparator)
  Interventions: Drug: Eptifibatide

INTERVENTIONS:
Drug: Eptifibatide — Intracoronary injection of Eptifibatide injected in two consecutive bolus of 180 mcg/kg each, followed immediately by continuous infusion of 2 mcg/kg/min for 12 hs.
  Arms: Eptifibatide (intracoronary)
Drug: Eptifibatide — Intravenous injection of Eptifibatide in two consecutive boluses of 180 mcg/kg followed by continuous intravenous injection dosing 2 mcg/kg/min for 12 hours
  Arms: Eptifibatide (intravenous)

SUMMARY:
The achievement of high local concentration of Eptifibatide, a GP 2b3a inhibitor,via direct intracoronary injection, promotes (in vitro) clot disaggregation. It remains unclear if it is of superior benefit than the routine intravenous administration of these agents.

In patients presenting with acute myocardial infarction, and undergoing primary coronary intervention, intracoronary administration of Eptifibatide may increase local drug concentration by several orders of magnitude and promote clot disaggregation with a minimal increase in systemic drug concentration, and in that way enhancing myocardial perfusion and survival.

DETAILED DESCRIPTION:
Patients will be randomized, prospectively, single blinded into one of two arms:1)intravenous administration of Eptifibatide and 2) intracoronary administration. The primary end-point will be the angiographic achievement of TIMI 3 flow at the infarct related artery and TIMI myocardial perfusion grade (blush) and the electrocardiographic surrogate of myocardial perfusion the ST segment resolution.

The secondary end-points will be the occurrence of bleeding or hemorrhagic complication according to TIMI classification and the LVEF at one month compared with baseline

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction candidate for primary coronary angioplasty, presenting within 12 hours of onset of pain and ability to clearly identified only one infarct related artery.

Exclusion Criteria:

* Contraindications for antiplatelet therapy such as bleeding disorders,
* Thrombocytopenia,
* Severe uncontrolled hypertension,
* Recent stroke (<6 months),
* Intracranial hemorrhage at any time
* Patients after recent major surgery (<30 days),
* Previous myocardial infarction
* Previous revascularization either by CABG or PCI and 9)patients presented with cardiogenic shock.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Coronary angiography | At the time of the procedure

SECONDARY OUTCOMES:
Electrocardiogram | 90 min after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Medical Center, Beer Yakov, Beer Yakov, Israel